CLINICAL TRIAL: NCT04207554
Title: Clinical Investigation for the Preview® hCG Urine/Serum Combo Pregnancy Test
Acronym: Preview® hCG
Status: Completed | Type: Observational
Sponsor: Guangzhou Wondfo Biotech Co., Ltd (Industry)
Collaborators: Nova Clinical Solutions, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: WF2019-01
Record Dates: First submitted 2019-12-18; First posted 2019-12-23 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Pregnancy
Keywords: Pregnancy; hCG; IVD; POCT

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Pregnancy Positive: Pregnant subjects within 11 weeks since the first day of last period.
  Interventions: Device: Test Device-Strip Format; Device: Test Device-Cassette Format; Device: Predicate Device
- Pregnancy Negative: Non-pregnant subjects.
  Interventions: Device: Test Device-Strip Format; Device: Test Device-Cassette Format; Device: Predicate Device

INTERVENTIONS:
Device: Test Device-Strip Format — Sponsor's investigational device
  Other Names: Preview® hCG Urine/Serum Combo Pregnancy Test-Strip Format
Device: Test Device-Cassette Format — Sponsor's investigational device
  Other Names: Preview® hCG Urine/Serum Combo Pregnancy Test-Cassette Format
Device: Predicate Device — Commercially available device
  Other Names: QuickVue+ hCG Combo Test

SUMMARY:
The objective of this study is to evaluate the agreement of the test device (Preview® hCG Urine/Serum Combo Pregnancy Test) with the predicate device, the QuickVue+ hCG Combo Test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult women of childbearing age.
* Who either request a pregnancy test, or require a pregnancy test for diagnostic studies or treatment.
* Signed and dated informed consent.

Exclusion Criteria:

* Minors.
* Adults who are unable to independently give consent for study.
* Known pregnancy (i.e. - patient appears obviously pregnant).
* Recent miscarriage or abortion and yet to have 2 complete menstrual cycles before study start.
* History of ectopic pregnancy, fibroids, congenital uterine anomaly that causes an irregular-shaped uterus.
* Taken any of the medications of contraceptives containing estrogen in last two weeks.
* Hemodynamically unstable.
* Moderately to severely ill-appearing or in moderate to severe pain.
* Technically not possible to obtain blood or urine from the study subject.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy adult women of childbearing age.
Study Population: The study will enroll healthy adult women of childbearing age.
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
Overall percent (%) agreement | 3 months
  The primary endpoint is the overall percent (%) agreement, which is the percentage of total subjects where the test (Preview® hCG Urine/Serum Combo Pregnancy Test) and the reference test (QuickVue+ hCG Combo Test) agree.

SECONDARY OUTCOMES:
Positive and negative percent agreement | 3 months
  The secondary endpoint is the positive percent agreement and negative percent agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Liu, Master, Study Chair — Guangzhou Wondfo Biotech Co., Ltd
Locations (6):
- United States (6):
  - National Insitute of Clinical Research, Garden Grove, California
  - National Research Institute-Huntington Park, Huntington Park, California
  - Downtown L.A. Research Center, Inc, Los Angeles, California
  - National Research Institute-Westlake, Los Angeles, California
  - National Research Institute-Panorama City, Panorama City, California
  - National Research Institute-Santa Ana, Santa Ana, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] WIDE L, GEMZELL CA. An immunological pregnancy test. Acta Endocrinol (Copenh). 1960 Oct;35:261-7. doi: 10.1530/acta.0.xxxv0261. No abstract available. PMID 13785019
- [Result] Batzer FR. Hormonal evaluation of early pregnancy. Fertil Steril. 1980 Jul;34(1):1-13. doi: 10.1016/s0015-0282(16)44829-6. No abstract available. PMID 6995156
- [Result] Braunstein GD, Rasor J, Danzer H, Adler D, Wade ME. Serum human chorionic gonadotropin levels throughout normal pregnancy. Am J Obstet Gynecol. 1976 Nov 15;126(6):678-81. doi: 10.1016/0002-9378(76)90518-4. PMID 984142
- [Result] Braunstein GD, Vaitukaitis JL, Carbone PP, Ross GT. Ectopic production of human chorionic gonadotrophin by neoplasms. Ann Intern Med. 1973 Jan;78(1):39-45. doi: 10.7326/0003-4819-78-1-39. No abstract available. PMID 4734160
- [Result] Catt KJ, Dufau ML, Vaitukaitis JL. Appearance of hCG in pregnancy plasma following the initiation of implantation of the blastocyst. J Clin Endocrinol Metab. 1975 Mar;40(3):537-40. doi: 10.1210/jcem-40-3-537. PMID 1117063
- [Result] Lenton EA, Neal LM, Sulaiman R. Plasma concentrations of human chorionic gonadotropin from the time of implantation until the second week of pregnancy. Fertil Steril. 1982 Jun;37(6):773-8. doi: 10.1016/s0015-0282(16)46337-5. PMID 7115557